CLINICAL TRIAL: NCT05787327
Title: Assessing the Efficacy and Safety of Yinqiaosan-Maxingganshitang in the Treatment of the Major Symptoms of Mild and Moderate COVID-19 by Telemedicine - a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: RCT for Yinqiaosan-Maxingganshitang in the Treatment of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID Acute study
Record Dates: First submitted 2023-03-23; First posted 2023-03-28 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ephedrae herba

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Yinqiaosan-Maxingganshitang ) (Experimental): Chinese Medicine granules
  Interventions: Drug: Chinese Herb
- Placebo (Placebo Comparator): Placebo granules
  Interventions: Diagnostic Test: Placebo

INTERVENTIONS:
Drug: Chinese Herb — Yinqiaosan-Maxingganshitang granules
  Other Names: CM
  Arms: Active treatment (Yinqiaosan-Maxingganshitang )
Diagnostic Test: Placebo — Placebo
  Other Names: Plavebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled clinical trial. This study is to evaluate the effectiveness and safety of Yinqiaosan-Maxingganshitang in the treatment of the major symptoms of mild and moderate COVID-19 patients by telemedicine.

DETAILED DESCRIPTION:
Subjects who are diagnosed with COVID-19 by RATs or PCR tests and fulfilled the eligibility criteria will receive a maximum of 14 days of treatment with Yinqiaosan-Maxingganshitang (with or without specified additions) or placebo and will be followed up on day 7, 14 and 35 after receiving medication (day 0).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years;
* Tested positive for COVID-19 by RATs, Deep Throat Saliva (DTS) or Throat/Nasal swab RT-PCR tests;
* Patient diagnosed with mild to moderate COVID-19 based on the "Coronavirus disease 2019 (COVID-19) Treatment Guidelines" published by National Institutes of Health;
* Duration of symptoms ≤ 72 hours (Start from the presence of the major symptoms of COVID-19: Fever: oral temperature >37.2°C, or cough score ≥2, or fatigue score ≥2);
* Diagnosed with pattern of wind and heat invading the surface and/or pattern of intense exuberance of lung heat by a registered Chinese medicine practitioner (CMP) (Diagnostic criteria are the corresponding criteria in the "Diagnosis standards for common syndromes in traditional Chinese medicine)" published by "Diagnostic Subcommittee of China Association of Traditional Chinese Medicine in 2008, with ≥20 as the threshold for determination);
* Explicit declaration of willingness to participate in the study at the time of videoconference screening after reading the electronic informed consent form (written consent form have to signed after inclusion).

Exclusion Criteria:

* Diagnosed of Asymptomatic or Presymptomatic Infection, Severe Illness or Critical Illness of COVID-19 based on the "Coronavirus disease 2019 (COVID-19) Treatment Guidelines" published by National Institutes of Health
* Known allergy to the Chinese medicines or other ingredients of the investigational medicinal products (IMP) used in this study;
* Known pregnancy or lactation;
* Known immunocompromised patient (such as malignancy, organ or bone marrow transplant, AIDS or low immune function caused by long-term use of corticosteroids or other immunosuppressants)
* Known obesity (Body Mass Index [BMI] ≥30)
* Heavy smoker (≥400 cigarettes/year)
* Known history of cardiovascular and cerebrovascular diseases (including hypertension), chronic lung disease (chronic obstructive pulmonary disease, moderate and severe asthma or interstitial lung disease), diabetes, chronic liver disease (ALT/AST ≥ 2× the upper limit of normal [ULN], Bilirubin-Total ≥ 1.5ULN), chronic kidney disease (Creatinine ≥1.5ULN), cancer or other chronic diseases.
* Known history of dysphagia or any gastrointestinal disorder that affects drug absorption (such as gastroesophageal reflux disease [GERD], chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, gastrectomy);
* Suspected or known history of alcohol or substance abuse or mental illness;
* Subjects having participated in other clinical studies in the past three months;
* Any other condition that in the opinion of the investigators could compromise the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Time for the body temperature to change to normal | From baseline to week 19
  The time between starting medication and body temperature dropping to normal (oral temperature ≤ 37.2℃ and maintain 24 hours).

SECONDARY OUTCOMES:
Time of negative Rapid Antigen Test | From baseline to reaching outcome
  2. The negative rate of Rapid Antigen Tests (RATs) at day 14 and the negative conversion time (two successive negative RATs result with at least 24 hours interval)
Remission rate of cough | 14 days
  The remission of cough will be measured by the score rating from 0 to 4, which representing "None", "Mild", "Moderate", "Severe" and "Very severe" respectively.
  The score of 1 or below and maintain for 24 hours will be counted as remission.
Remission rate of fatigue | 14 days
  The remission of fatigue will be measured by the score rating from 0 to 4, which representing "None", "Mild", "Moderate", "Severe" and "Very severe" respectively.
  The score of 1 or below and maintain for 24 hours will be counted as remission.
Time of remission of cough | From baseline to week 19
  Time from the start of treatment to the symptom remission
Time of remission of fatigue | From baseline to week 19
  Time from the start of treatment to the symptom remission
Disappearance rate of COVID symptom | 14 days
  The disappearance rate of the COVID symptom
Incidence to severe illness | From baseline to 19 weeks
  Incidence of the progression to severe ot critical illness during the trial
Mortality | 21 days
  All-cause mortality at the 21th days after stopping the medications
Utilization rate of rescue drugs | 14 days
  Utilization rate of antipyretic, Paxlovid and molnupiravir within 14 days
Dosage of rescue drugs | 14 days
  Dosage of antipyretic, Paxlovid and molnupiravir within 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- Hong Kong Institute of Integrative Medicine, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Sum CH, Li TW, Zhang H, Hung HY, Fong BYF, Lin WL, Chow TY, Leung KC, Lo CW, Chia CP, Chan KL, Lin ZX. Assessing the efficacy and safety of Yinqiao powder-maxing Ganshi decoction in the treatment of the major symptoms of mild and moderate COVID-19 by telemedicine-study protocol for a randomized, double-blind, placebo-controlled trial. Front Pharmacol. 2024 Jan 8;14:1261338. doi: 10.3389/fphar.2023.1261338. eCollection 2023. PMID 38259270